CLINICAL TRIAL: NCT04622111
Title: One Centre, Single Ascending Dose and Double Blind Multiple Ascending Dose, Safety and Pharmacokinetics Phase I Study of CPL207280 Compound in Healthy Volunteers.
Brief Title: Safety and Pharmacokinetics Study of CPL207280 Compound in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 01GPR2019
Record Dates: First submitted 2020-11-06; First posted 2020-11-09 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — CPL207280; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only PART B will be double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPL207280 (Experimental): PART A: 8 cohorts are to receive single dose of IMP.Each participant is to take single dose of IMP. There is to be dose escalation between cohorts.
  PART B: 4 cohorts are to receive multiple dose of IMP. Each participant is to take IMP once daily for 14 days. There is to be dose escalation between cohorts.
  Interventions: Drug: CPL207280
- Placebo (Placebo Comparator): PART B: 2 Participants from each of 4 cohorts (total of 8 participants) are to receive masking placebo tablet once daily for 14 days. There is to be dose escalation between cohorts. Participants are to be randomized within cohorts.
  Interventions: Drug: Placebo
- CPL207280 120 mg + Metformin 750 mg (Experimental): 1 cohort (total of 12 participants) are to receive single dose of IMP in fed and fasted state, IMP with metformin and metformin alone to assess the effect of food and metformin on bioavailability of CPL207280. There is to be one week wash-out between four treatments periods for this cohort.
  Interventions: Drug: CPL207280; Drug: Metformin hydrochloride 750 mg

INTERVENTIONS:
Drug: CPL207280 — IMP is a tablet with CPL207280 as an Active Pharmaceutical Ingredient (API).
  Arms: CPL207280; CPL207280 120 mg + Metformin 750 mg
Drug: Placebo — matching placebo tablet
  Arms: Placebo
Drug: Metformin hydrochloride 750 mg — IMP is a tablet with Metformin hydrochloride as an Active Pharmaceutical Ingredient (API).
  Other Names: Glucophage XR 750 mg
  Arms: CPL207280 120 mg + Metformin 750 mg

SUMMARY:
The planned study is to determine the safety and pharmacokinetic properties of CPL207280 compound after single and multiple (two weeks) administration in healthy volunteers.

DETAILED DESCRIPTION:
This is to be one-centre, single ascending dose and double-blind multiple ascending dose two part study of CPL207280 compound in healthy volunteers. PART A is a single dose, open-label part with CPL207280 compound administered with dose escalation between cohorts.Additionaly assessing the effect of food and effect of metformin on bioavailability of CPL207280 is to be done in additional cohort. PART B is a multiple, double-blind part with CPL207280 compound administered for 14 days with dose escalation between cohorts. Participants in this part are to be randomized to receive Investigational Medicinal Product (IMP) or placebo in 3:1 ratio. Safety and pharmacokinetic properties of CPL207280 compound is to be determined following different doses in single oral IMP administration in PART A and different doses of IMP administered orally for two weeks in PART B.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female or male
* Body-mass index (BMI): ≥ 18.5 kg/m² and < 29.9 kg/m²,
* Physical examination without any clinically relevant abnormality,
* Clinical laboratory results in hematology or renal/hepatic test and clinical laboratory results in other tests without any clinically relevant abnormalities as assessed by Investigator,
* Non-smoker and non-user of tobacco products for at least 3 months before screening,
* Subject able to provide written informed consent after receiving information about the trial,
* Informed Consent Form signed and dated prior to Screening evaluations,
* Ability and willingness to comply with the requirements of the study protocol,
* Volunteer (or his/her partner) of childbearing potential willingness to use acceptable forms of contraception.

Exclusion Criteria:

* Known allergy, hypersensitivity, intolerance or contraindication to other drugs similar in structure or class to CPL207280 compound, or to any excipients of the formulation,
* Any known significant current or past acute or chronic disease or condition of the: circulatory, respiratory, hematopoietic, endocrine, nervous and musculoskeletal system, alimentary and urinary tracts, allergic disease, genetic or psychiatric disorder that could influence the present general health condition, at the Investigator's discretion,
* A long QT interval analysis syndrome (in the interview) or is under the treatment with antiarrhythmic drugs,
* Current disease of the alimentary tract, liver or kidneys that may influence absorption, distribution and/or elimination of the studied drug, as assessed by the Investigator and documented in the medical history,
* Medical condition that requires administration of other drugs or use of any drug within the 4 weeks preceding the first IMP administration and during the entire study. Drugs commonly used with fast metabolism may be administered and is up to Investigator discretion (i.e. pain killers),
* Participation in other clinical trials, where at least one dose of study drug was administered, within 90 days preceding the screening phase,
* Blood drawn within 30 days prior to inclusion in this study (more or equal to 300 mL),
* Positive results from pregnancy test in female volunteers,
* Lactation in female volunteers,
* Hypotension or hypertension in medical history,
* Narcotic and alcohol addiction or abuse,
* Positive results of HBsAg, anti-HCV or anti-HIV tests,
* Positive drug screen or alcohol breath tests,
* Subjects who adhere to a special diet (e.g. low calories, vegetarian,etc.).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) or administration of the maximum dose provided in the protocol after single and multiple oral administration of IMP. | up to 48 hours after single administration of IMP in PART A and up to 48 hours after the last IMP administration in PART B
  MTD is defined as the highest dose for which no more than 1 of the 6 treated volunteers (less than 1/3) exhibits dose limiting toxicity (DLT).
Safety and tolerability of IMP after single and multiple oral administration | up to 14 days in PART A and up to 28 days in PART B of the study
  Participants during hospitalization are to be closely observed to assure maximal safety and to collect occurrence of all adverse event. To follow-up on all study participants telephone calls with a request for information regarding their health condition are to be made.

SECONDARY OUTCOMES:
Cmax - maximum plasma concentration | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  The maximum concentration of the CPL207280 compound in plasma after IMP administration, obtained directly from the measured concentrations.
AUC(0-48) - area under the plasma concentration - time curve from time 0 to 48h after IMP administration | up to 48 hours after administration of IMP in PART A and after the IMP administration determined on Day 14 in PART B
  The AUC(0-48) is a measure of total plasma exposure to the drug from time point zero to 48 hours after IMP administration
AUC(0-24) - area under the plasma concentration - time curve from time 0 to 24h after IMP administration | up to 24 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1 and 8 in PART B
  The AUC(0-24) is a measure of total plasma exposure to the drug from time point zero to 24 hours after IMP
AUC(0-inf) - area under the plasma concentration - time curve from time 0 to infinity time | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  The AUC(0-inf) is a measure of total plasma exposure to the drug from time point zero extrapolated to infinity.
Tmax - time to reach maximum concentration | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  The Tmax is time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times.
Kel - terminal elimination rate constant | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  Kel is to be estimated via linear regression of time versus log of concentration.
T1/2 - The plasma elimination half-life | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  T1/2 is to be calculated as 0.693/Kel.
C (1,t) - CPL207280 concentration | Determined on Day 2, 3, 4, 5, 6, 7, 9, 10, 11, 12 and 13 in PART B
  The concentration of CPL207280 on day t before product administration.
C (Tmax, t) - CPL207280 concentration | Determined on Day 2, 3, 4, 5, 6, 7, 9, 10, 11, 12 and 13 in PART B
  The concentration on day t measured on time Tmax which was calculated in PART A of the study.
Glucose AUEC -area under the effect-time curve after IMP administration | up to 6 hours after administration of IMP in PART A and up to 6 hours after the IMP administration determined on Day 1, 8,14 in PART B
  The AUEC is a measure of total glucose concentration from time point zero to 6 hours after IMP
Insulin AUEC -area under the effect-time curve after IMP administration | up to 6 hours after administration of IMP in PART A and up to 6 hours after the IMP administration determined on Day 1, 8,14 in PART B
  The AUEC is a measure of total insulin concentration from time point zero to 6 hours after IMP
Proinsulin AUEC -area under the effect-time curve after IMP administration | up to 6 hours after administration of IMP in PART A and up to 6 hours after the IMP administration determined on Day 1, 8,14 in PART B
  The AUEC is a measure of total proinsulin concentration from time point zero to 6 hours after IMP
C-peptide AUEC -area under the effect-time curve after IMP administration | up to 6 hours after administration of IMP in PART A and up to 6 hours after the IMP administration determined on Day 1, 8,14 in PART B
  The AUEC is a measure of total c-peptide concentration from time point zero to 6 hours after IMP
Glucagon AUEC -area under the effect-time curve after IMP administration | up to 6 hours after administration of IMP in PART A and up to 6 hours after the IMP administration determined on Day 1, 8,14 in PART B
  The AUEC is a measure of total glucagon concentration from time point zero to 6 hours after IMP
AUC(0-tau, t)- area under the curve of plasma concentration vs time, from time point zero up to the time of 24h in day t | up to 24 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 and 14 in PART B
  AUC(0-tau, t) will be calculated according to the linear trapezoidal rule
Cav,t, averate IMP concentration on day t | up to 24 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 and 14 in PART B
  Cav,t, will be calculated as AUC(0-tau, t)/24h.
Fluctuation | up to 24 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 and 14 in PART B
  Fluctuation will be calcilated as a difference between C(Tmax,t) and C(1,t) relative to the Cav,t, calculated as (C(Tmax,t)-C(1,t))/Cav,t x 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- BioResearch Group Sp. z o.o., Kajetany, Nadarzyn, Poland

REFERENCES:
- [Derived] Bazydlo-Guzenda K, Buda P, Matloka M, Mach M, Stelmach F, Dzida R, Smuga D, Hucz-Kalitowska J, Teska-Kaminska M, Vialichka V, Dubiel K, Kaminska B, Wieczorek M, Pieczykolan J. CPL207280, a Novel G Protein-Coupled Receptor 40/Free Fatty Acid Receptor 1-Specific Agonist, Shows a Favorable Safety Profile and Exerts Antidiabetic Effects in Type 2 Diabetic Animals. Mol Pharmacol. 2021 Oct;100(4):335-347. doi: 10.1124/molpharm.121.000260. Epub 2021 Aug 4. PMID 34349026